CLINICAL TRIAL: NCT04860856
Title: Efficacy of Hematoma Block on Postoperative Pain After Femoral Intramedullary Rodding: A Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Ruixian Yue, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OS19011 IRB 2019-0366
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Femur Fracture
Keywords: Femoral Intramedullary Rod; Hematoma Block
MeSH Terms: conditions — Femoral Fractures | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Blinded, randomized control trial
Who Masked: Participant, Care Provider
Masking Description: The patients and the nursing staff who assess postoperative pain will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hematoma block (Experimental): Fracture site injection of 20 mL of 0.5% ropivacaine with an 18-gauge needle (150 mm length).
  Interventions: Drug: 0.5% ropivacaine
- Normal saline injection (Placebo Comparator): Fracture site injection of 20ml of normal saline.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: 0.5% ropivacaine — The maximal single dose of ropivacaine without vasoconstrictor is 2-3 mg/kg.9 0.5% ropivacaine has 5 mg/mL of ropivacaine. 20 mL of 0.5% ropivacaine has 100 mg of ropivacaine. 100 mg of ropivacaine can be toxic to a patient less than 33-50 kg or 73-110 lb. If a patient weighs less than 110 lb, the ropivacaine dose will be scaled down below 2 mg/kg.
  Arms: Hematoma block
Drug: Normal Saline — 20ml of normal saline
  Arms: Normal saline injection

SUMMARY:
The purpose of this study is to evaluate the efficacy of an intra-operative, post-fixation fracture hematoma block compared to saline control on postoperative pain control in patients with acute femoral shaft fractures. Our primary outcome measure is visual analog scale (VAS) pain scores which are recorded at regular intervals.

DETAILED DESCRIPTION:
This blinded, randomized control trial is being performed at the University of Cincinnati Medical Center.

Patients will be randomly assigned to one of two treatment groups: Group One will be comprised of patients treated with fracture site injection containing 20 mL of 0.5% ropivacaine with an 18-gauge needle (150 mm length), Group Two will be comprised of patients treated with fracture site injection containing 20ml of normal saline. The injection will be administered by the orthopaedic trauma team after the insertion of the final intramedullary implant and skin closure prior to final surgical dressing application. The injection will be performed in a standard fashion with aspiration of hematoma followed by the injection. All postoperative management will be per standard of care.

The size of the hematoma will have no effect on the procedure. When a hematoma block is utilized in the care of orthopaedic trauma patients, its aim is to infiltrate the anesthetic to the fracture edges and injured soft tissue to allow for pain control and fracture manipulation without additional sedation. Aspiration of the hematoma tells the clinician that the tip of the needle is near the fracture site and not in a neurovascular structure.

The maximal single dose of ropivacaine without vasoconstrictor is 2-3 mg/kg.9 0.5% ropivacaine has 5 mg/mL of ropivacaine. 20 mL of 0.5% ropivacaine has 100 mg of ropivacaine. 100 mg of ropivacaine can be toxic to a patient less than 33-50 kg or 73-110 lb. If a patient weighs less than 110 lb, the ropivacaine dose will be scaled down below 2 mg/kg.

Regional anesthesia including nerve blocks is not routinely used in the setting of traumatic femoral shaft fractures. A nerve block would compromise the patient's neurologic examination in the immediate postoperative period.

Randomization will be performed via Microsoft Excel to generate random numbers. Allocation will be concealed and revealed to the surgical team in the hour prior to the procedure. The patients and the nursing staff who assess postoperative pain will be blinded to the treatment allocation.

An a priori power analysis was performed to determine the sample size for the primary outcome measure. Prior literature has indicated that a difference of 1.3 on a VAS is clinically significant.5 Therefore, it was determined that a total of 44 patients were necessary per group to detect a 1.5-point difference on the VAS (power = 80%, p = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient at the University of Cincinnati Medical Center
* Skeletally mature patients
* Have an isolated, closed, acute traumatic femoral shaft fracture to be treated with a closed reduction and reamed intramedullary rod fixation

Exclusion Criteria:

* Unable to provide informed consent
* Member of a vulnerable patient population
* Have additional injuries
* Have a history of prior existing narcotic use or chronic pain management issues on presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-08-17 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain at 72 hours | Measured at 0, 8, 16, 24, 36, 48, and 72 hours postoperatively
  Postoperative pain will be assessed using a visual analog scale

SECONDARY OUTCOMES:
Narcotic usage | Narcotic usage will be assessed through 72 hours postoperatively
  Oral morphine equivalents will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: He C S, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alioto RJ, Furia JP, Marquardt JD. Hematoma block for ankle fractures: a safe and efficacious technique for manipulations. J Orthop Trauma. 1995 Apr;9(2):113-6. doi: 10.1097/00005131-199504000-00004. PMID 7776029
- [Background] Bear DM, Friel NA, Lupo CL, Pitetti R, Ward WT. Hematoma block versus sedation for the reduction of distal radius fractures in children. J Hand Surg Am. 2015 Jan;40(1):57-61. doi: 10.1016/j.jhsa.2014.08.039. Epub 2014 Oct 11. PMID 25306504
- [Background] Case RD. Haematoma block--a safe method of reducing Colles' fractures. Injury. 1985 Jul;16(7):469-70. doi: 10.1016/0020-1383(85)90168-8. PMID 4030071
- [Background] Herrera JA, Wall EJ, Foad SL. Hematoma block reduces narcotic pain medication after femoral elastic nailing in children. J Pediatr Orthop. 2004 May-Jun;24(3):254-6. doi: 10.1097/00004694-200405000-00003. PMID 15105718
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Koehler D, Marsh JL, Karam M, Fruehling C, Willey M. Efficacy of Surgical-Site, Multimodal Drug Injection Following Operative Management of Femoral Fractures: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Mar 15;99(6):512-519. doi: 10.2106/JBJS.16.00733. PMID 28291185
- [Background] Johnson PQ, Noffsinger MA. Hematoma block of distal forearm fractures. Is it safe? Orthop Rev. 1991 Nov;20(11):977-9. PMID 1749663
- [Background] Dimopoulou I, Anagnostou TL, Prassinos NN, Savvas I, Patsikas M. Effect of intrafragmentary bupivacaine (haematoma block) on analgesic requirements in dogs undergoing fracture repair. Vet Anaesth Analg. 2017 Sep;44(5):1189-1197. doi: 10.1016/j.vaa.2017.01.005. Epub 2017 Mar 6. PMID 29100681
- [Derived] Yue RA, Shah NS, Matar RN, Sagi HC. Efficacy of Hematoma Block After Intramedullary Rod Fixation of Femoral Shaft Fractures: A Prospective, Double-Blinded, Randomized Controlled Trial. J Orthop Trauma. 2023 Sep 1;37(9):429-432. doi: 10.1097/BOT.0000000000002623. PMID 37199424